CLINICAL TRIAL: NCT01097928
Title: Pulmonary Embolism Response to Fragmentation, Embolectomy, & Catheter Thrombolysis: The PERFECT Registry
Brief Title: Pulmonary Embolism Response to Fragmentation, Embolectomy, & Catheter Thrombolysis: PERFECT
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Adventist Midwest Health (Unknown); Weill Medical College of Cornell University (Other); Memorial Hospital of South Bend (Other); Northside Hospital, Inc. (Other); Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, William Kuo, Professor - Interventional Radiology, Stanford University
Other Study IDs: SU-03292010-5502; eProtocol ID 14793
Record Dates: First submitted 2010-03-30; First posted 2010-04-02 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients undergoing Pulmonary Embolectomy
  Interventions: Procedure: Catheter directed debulking of Pulmonary Embolus

INTERVENTIONS:
Procedure: Catheter directed debulking of Pulmonary Embolus — A catheter will be used to break up the pulmonary embolism

SUMMARY:
A prospective observational study to evaluate the safety and effectiveness data of catheter-directed therapy (CDT) including percutaneous mechanical thrombectomy (PMT) for treatment of acute pulmonary embolism (PE)

DETAILED DESCRIPTION:
The primary objective of this study is to capture high quality patient safety and effectiveness data on CDT for acute PE. The goal will be achieved by capturing a concise set of immediate and short-term functional and clinical outcome data for PE patients undergoing CDT.

Secondary study objectives include the following:

- To assess and benchmark clinical practice patterns (patient selection, optimal technique, use of procedure worldwide)

These objectives will be achieved through the capture of selected process data for patients included in the registry. Data collected in this study may also be used to develop and refine standards of care for use of CDT for PE and to facilitate the design of randomized clinical trials

ELIGIBILITY:
Inclusion Criteria:

* Must be Age greater than or equal to 18
* Obtain informed written consent.
* Diagnosed with acute pulmonary embolism (PE) (< 14 days)
* Catheter-directed therapy (CDT) was performed to treat acute PE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient who has developed a pulmonary embolism, and who will be undergoing catheter directed debulking of the embolus.
Sampling Method: Non-Probability Sample
Enrollment: 333 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Resolution of hypoxia | Post-procedure and 3 months
Survival from acute PE | Post-procedure and 3 months
Stabilization of hemodynamics | Post-procedure and 3 months

SECONDARY OUTCOMES:
Clinical practice patterns across centers | 5yrs

CONTACTS AND LOCATIONS:
Overall Officials: William T Kuo MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Kuo WT, Banerjee A, Kim PS, DeMarco FJ Jr, Levy JR, Facchini FR, Unver K, Bertini MJ, Sista AK, Hall MJ, Rosenberg JK, De Gregorio MA. Pulmonary Embolism Response to Fragmentation, Embolectomy, and Catheter Thrombolysis (PERFECT): Initial Results From a Prospective Multicenter Registry. Chest. 2015 Sep;148(3):667-673. doi: 10.1378/chest.15-0119. PMID 25856269